CLINICAL TRIAL: NCT00615576
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SB-656933 Following 14 Days Repeat Dosing in Healthy Male Smokers
Brief Title: Repeat Dose Study in Male Healthy Volunteer Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CR2111256
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Smoker,; Male,; Chronic Obstructive Lung Disease; Cystic Fibrosis,; Healthy Volunteer,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis | interventions — SB 656933

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving SB-656933 (Experimental): Eligible subjects will be randomized to receive once daily doses of 100 milligrams of SB- 656933 for 14 days.
  Interventions: Drug: SB-656933
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will be randomized to receive placebo for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB-656933 — SB-656933 will be available as white film coated, round tablet and will be available in strengths of 50 milligrams, administered orally once daily.
  Arms: Subjects receiving SB-656933
Drug: Placebo — A placebo tablet to visually match the SB-656933 tablet will also be supplied, administered orally once daily.
  Arms: Subjects receiving placebo

SUMMARY:
This is a 4 to 6 week study to look at the safety and PK profile of SB656933 in healthy male smokers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male smokers who are between 18-65 years of age with normal genitourinary anatomy based on physical examination.
* The subjects should have a normal colour Doppler epididymal ultrasound (normal blood flow and epididymal morphology) at screening.
* The first 10 mL of urine voided (VB1) should be normal at screening and pre-dose.
* Male subjects must agree to abstain from or use a condom during sexual intercourse with pregnant females; or use a condom/spermicide, in addition to having their female partner use another form of contraception, such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of the first dose of study medication until 84 days after the last dose of study medication.
* The subject has a QTc(B) <450msec at screening or prior to dosing
* Body weight = 50 kg (110 pounds) and body mass index (BMI) between 19 and 30 inclusive where: BMI =weight in kg/(height in meters)2
* Healthy male smokers must smoke more than 10 cigarettes per day, for at least 2 months prior to screening and less than 30 cigarettes per day at the time of enrolment.
* Subjects with Forced Expiratory Volume (FEV1)=80% predicted and FEV1/Forced Vital Capacity (FVC) ratio=0.7.
* Signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or 12-lead ECG.
* The subject has liver function tests (LFT) elevated above the reference range at pre-study screening that remain elevated with a repeat LFT (to be discussed with the sponsor, if necessary).
* Subjects with absolute neutrophil count (ANC) = 2.0x109/L.
* Subjects who have previously been exposed to testicular radiotherapy.
* Subjects who have had previous testicular or prostate surgery including vasectomy.
* History of prostatitis, epididymitis, epididymal cysts, structural abnormalities or testicular cancer.
* Subjects with abnormalities of the renal tract, renal stones or history of Urinary Tract Infections (UTI's).
* Positive drug or alcohol test at screening or prior to dosing.
* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody at screening
* Use of prescription or non-prescription medication in the last 7 days or 5 half-lives (whichever is longer) , particularly drugs that are P450 CYP3A4, CYP2B6, CYP2C8 or OATP1B1 substrates with a narrow therapeutic index , and including vitamins and herbal remedies such as St John's Wort prior to dose of study medication.
* Consumption of grapefruit or grapefruit juice within seven days prior to the first dose of study medication.
* Donation of blood in excess of 500 mL within a 56 day period prior to dosing.
* Exposure to more than 3 new chemical entities within 12 months prior to the first dosing day.
* Participation in a trial with any drug within 3 months before the start of the study or participation in a trial with a new chemical entity within 4 months before the start of the study.
* Are receiving treatment for smoking cessation.
* Are using tobacco products other than cigarettes (e.g. pipes, cigars, snuff, chewing tobacco).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03-26 (Actual); Primary Completion 2008-07-24 (Actual); Study Completion 2008-07-24 (Actual)

PRIMARY OUTCOMES:
-what the body does to the drug over a 17 day of dosing with 100mg of SB656933. -Safety of SB-656933: Adverse events, blood pressure, heart rate, electrocardiogram, epididymal ultrasound and lab tests | 17 days
-what the body does to the drug over a 17 day of dosing with 100mg of SB656933 by taking PK samples at: | pre-dose and at 0.5,1,2,3,4,6,8,12 and 24 hours post-dose on days 1 and 14; pre-dose on Day7. Additional samples at 32, 48 and 72 hours post-dose wil
-Safety of SB-656933: Adverse events every day for entire study period: blood pressure , heart rate and temperature | taken pre-dose, 30min, 1hr, and 2hr on Day1, Day2, Day7 and Day14 (supine only);
electrocardiogram | pre-dose, 2hr and 4 hr on Day1

SECONDARY OUTCOMES:
- Looking at the actual sample size data to determine a larger theoretical population. -What the drug does to the body when present at its lowest level on day 14 as compared before drug given. | 17 days
Safety and tolerability of SB-656933 in subjects with cystic fibrosis, including adverse events, vital signs, clinical laboratory assessments, electrocardiographic (ECG) parameters, and lung function (FVC, FEV1) | Up to Day 28
Fluorocytometric quantitation of CXCL1-induced CD11b expression on peripheral blood neutrophils in ex-vivo assay. | Up to Day 14
Neutrophil shape change in response to stimulation with CXCL-1 in whole blood ex-vivo gated autofluorescence forward scatter (GAFS) assay. | Up to Day 14
Looking at the actual sample size data to determine a larger theoretical population. | Up to Day 14
What the drug does to the body when present at its lowest level on day 14 as compared before drug given. | on day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study CR2111256 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CR2111256?search=study&study_ids=CR2111256#rs